CLINICAL TRIAL: NCT05340920
Title: Relevance of Sensitization to Fenugreek in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Amandine DIVARET-CHAUVEAU, Head of pediatric allergy department, Central Hospital, Nancy, France
Other Study IDs: 2021PI211
Record Dates: First submitted 2022-04-08; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Allergy to Fenugreek
Keywords: allergy; children; legumes; sensitization; diagnostic
MeSH Terms: conditions — Hypersensitivity; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Oral Food Challenge — diagnostic values of skin prick test and specific IgE for allergy confirmed by oral food challenge (routine, not an intervention)

SUMMARY:
The prevalence of allergy to legumes is inscreasing, especially in children and for some of these legumes, little is known and there are not included in the list of priority allergen. The overall goal of this study is to improve knowledge about fenugreek allergy. The principal aim is to evaluate the prevalence of allergy to fenugreek confirmed by a positive oral food challenge in children sensitized to fenugreek. The secondary objectives are to describe the case of allergy to fenugreek (co-allergies, severity, age..), to evaluate diagnostic values of skin prick-tests and specific IgE and to compare the molecular profile of specific IgE to peanut between sensitization to fenugreek without allergy and sensitization with a confirmed allergy

ELIGIBILITY:
Inclusion Criteria:

* Children for whom an oral food challenge to fenugreek has been performed between the 1st January 2017 and the 15th April 2022 and for whom skin prick test and/or specific IgE to fenugreek are avalaible

Exclusion Criteria:

* patient over 18 years old
* undeterminate oral food challenge

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged from 1 to 17 years old, sensitized to fenugreek with an evaluation of their tolerance to fenugreek by an oral food challenge
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Oral food challenge to fenugreek | 2017-2022
  Astier's score 0 to 4 (0=negative, 1 and 2=mild to moderate reaction, 3 and 4 = severe reaction)
skin prick-test to fenugreek | 2017-2022
  skin prick test positive if wheal size superior to 3mm
specific IgE to fenugreek | 2017-2022
  specific IgE positive if value superior to 0.35kU/L

SECONDARY OUTCOMES:
severity of allergy | 2017-2022
  reactogenic dose (from 1 to 1000mg of fenugreek)
molecular profile for peanut allergy | 2017-2022
  IgE values for rAra h1, h2, h3, h6, h8, h9

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Divaret-Chauveau, MD, Principal Investigator — centre hospitalo-universitaire de Nancy
Locations (1):
- Centre Hospitalo-Universitaire de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No